CLINICAL TRIAL: NCT01305083
Title: A Randomized, Double Blind, Placebo Controlled, Multicentric Study to Assess the Efficacy and Safety of Udenafil Tablets in Patients Suffering From Erectile Dysfunction.
Brief Title: Efficacy and Safety Study of Udenafil Tablets in Erectile Dysfunction.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abdi Ibrahim Ilac San. ve Tic A.S. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AI2010-01
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — udenafil

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Udenafil (Active Comparator): Active Ingredient
  Interventions: Drug: Udenafil; Drug: Placebo
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Udenafil; Drug: Placebo

INTERVENTIONS:
Drug: Udenafil — Placebo-control
Drug: Placebo — Placebo

SUMMARY:
This randomized, double blind, placebo controlled, multicentric, clinical study will assess the efficacy and safety of Udenafil (100 mg) tablets in patients suffering from erectile dysfunction(ED).

ELIGIBILITY:
Inclusion Criteria:

* Male patients of 18 to 60 years of age.
* Patients in a stable, monogamous sexual relationship with a female partner for at least 6 months and willing to maintain this relationship for the duration of the study.
* Patients with established diagnosis of erectile dysfunction (ED) of organic, psychogenic or mixed etiology for at least 6 months duration.
* Patient willing to attempt at least one sexual intercourse in a week for the entire treatment.

Exclusion Criteria:

* Patients with total erectile failure or any other sexual disorder such as hypoactive sexual desire.
* Patients who have previously failed to respond to PDE-5 inhibitors like Sildenafil, Vardenafil or Tadalafil.
* Patients who have used other erectile dysfunction therapies within 14 days (2 weeks) prior to entering into this study (i.e. visit 1).
* Patients with hypogonadism or anatomical deformity of the penis such as severe penile fibrosis or Peyronie's disease or penile trauma.
* Patients with a history of major psychiatric disorder.
* Patients with a history of significant pathological cardiovascular conditions such as: congestive heart failure, life-threatening arrhythmia or ischemic heart disease within the past 6 months.
* Patients with a history of central nervous system disorders such as stroke, transient ischemic attacks or spinal cord injury or a radical prostatectomy or radical pelvic surgery.
* Patients with hypotension (<90/50) or uncontrolled hypertension (>170/100), uncontrolled diabetes, hepatic impairment (SGOT or SGPT levels > 3 x Upper Normal Limit), renal impairment (serum creatinine > 2.5mg/dl), hematological disorders such as bleeding disorders.
* Patients with a history of retinitis pigmentosa, proliferative diabetic retinopathy or non-arteritic anterior ischemic optic neuropathy (NAION).
* Patients with a history of sickle cell disease, multiple myeloma, leukemia or any other disorders that may cause priapism.
* Patients on concomitant treatment with nitrates/nitrites(NO) donor, CYP3A4 inhibitors, CYP3A4 inducers, anticoagulants, androgens, antiandrogens or trazodone.
* Patients with known hypersensitivity to PDE 5 inhibitors like Sildenafil, Vardenafil or Tadalafil.
* Patient with known diagnosis to AIDS or with a positive HIV result at study screening visit.
* Patients with any other serious concurrent illness or malignancy.
* Patients with continuing history of alcohol and / or drug abuse.
* Participation in another clinical trial in the past 30days.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
IIEF | 8 week

SECONDARY OUTCOMES:
Changes in the total score of IIEF at the end of the treatment compared to baseline. | 8 week
Changes in score of Question 3 (SEP2) and Question 4 (SEP3) of IIEF questionnaire at the end of the treatment period as compared to baseline. | 8 week
Overall assessment of efficacy (GAQ) to the study medication at the end of the study. | 8 week

CONTACTS AND LOCATIONS:
Locations (4):
- Turkey (Türkiye) (4):
  - Ankara
  - Istanbul
  - Izmir
  - Mersin